CLINICAL TRIAL: NCT07167823
Title: The Role of Decortication in Complex Empyema Cases: Multidrug Resistance and Tuberculosis at the Forefront
Status: Completed | Type: Observational
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Principle Investigator, University of Health Sciences Lahore
Other Study IDs: IRB/2025/1546/SIMS
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pleural Empyema; Tuberculosis (TB); Bacterial Sepsis
Keywords: Multi-drug resistance; Decortication; Bacterial empyema thoracis; tuberculous empyema thoracis
MeSH Terms: conditions — Empyema, Pleural; Tuberculosis | interventions — Cerebral Decortication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bacterial empyema thoracis: all participants that were diagnosed as having empyema thoracis due to bacterial organisms, also included multi-drug resistant organisms.
  Interventions: Procedure: Decortication
- Tuberculous Empyema Thoracis: all participants that were diagnosed as having empyema thoracis due to mycobacterium tuberculosis, also included multi-drug resistant organisms.
  Interventions: Procedure: Decortication

INTERVENTIONS:
Procedure: Decortication — removal of fibrinous infected material from pleural cavity and thick fibrous entrapping peel over the lung resulting in full expansion of lung.
  Groups: Bacterial empyema thoracis
Procedure: Decortication — removal of fibrinous infected material and thick fibrinous entrapping peel over the lung
  Groups: Tuberculous Empyema Thoracis

SUMMARY:
Empyema is a problem that thoracic surgeons deal in everyday practice. The main goal of treatment is evacuating the pus and fibrin deposits in the thoracic cavity for complete lung expansion. This study aims to report a detailed microbiological profile of patients operated for empyema thoracis and also correlate it with perioperative clinical outcomes. Patients who underwent surgery for empyema thoracis between January 2022 to June 2025 were included in the study. This study was carried out at two centers; Thoracic Surgery Department, Services Hospital Lahore. Patients were taken up for surgery after thorough preoperative evaluation. Perioperative outcomes were correlated with the results of microbiological analysis to evaluate their effect on clinical outcomes. This study highlights the emergence of Gram-negative organisms in bacterial empyema and emergence of multidrug resistance in tubercular empyema. Clinical outcome correlation revealed increased complications in culture-positive cases in both tubercular and nontubercular empyemas

DETAILED DESCRIPTION:
Pleural empyema, defined as the accumulation of infected pleural fluid, remains a significant clinical challenge globally despite advancements in medical and surgical therapies. In the United States, approximately 32,000 cases of pleural empyema are diagnosed annually , with mortality rates ranging from 5% to 20%. In Pakistan, though national data is lacking, the burden is presumed to be disproportionately higher due to the high prevalence of tuberculosis (TB) and the rising threat of multidrug resistance (MDR). This dual burden necessitates the adoption of robust, evidence-based strategies tailored to the healthcare challenges of the region.

Effective management of empyema requires a multidisciplinary approach involving thoracic surgeons, pulmonologists, infectious disease specialists, and microbiologists. While the initial management focuses on prompt antibiotic therapy and drainage of infected pleural fluid, the emergence of MDR bacterial pathogens and TB-specific challenges complicate the treatment landscape. In particular, MDR bacterial empyemas often demand susceptibility-guided antibiotic regimens, while tuberculous empyemas are complicated by delays in diagnosis and the increasing prevalence of MDR-TB. The intersection of these issues makes individualized management strategies essential in countries like Pakistan, where TB remains a major public health concern.

Surgical intervention is a cornerstone in the management of complicated or refractory empyema, with decortication being the gold-standard procedure to restore lung expansion and achieve definitive source control. At our tertiary care thoracic surgery center, approximately 30-40% of empyema cases require escalation to surgical decortication, consistent with global trends. Both thoracoscopic and open approaches are utilized depending on the stage of the disease and patient-specific factors. Surgical outcomes, however, are influenced by the underlying microbiological profile, as highlighted by a study involving 285 operated cases of empyema thoracis and reported that 58.2% of cases were tubercular in origin, with a mycobacterial culture positivity rate of 19.28%, of which 21.8% were MDR. Nontubercular cases, accounting for 41.8%, were predominantly caused by Gram-negative organisms, with Pseudomonas aeruginosa being the most frequent isolate. These findings align with the microbiological trends observed in our practice, where both MDR pathogens and TB complicate clinical decision-making.

Postoperative management, particularly the duration of antibiotic therapy following decortication, remains a contentious issue with significant variability in global guidelines. The British Thoracic Society recommends a minimum of three weeks of antibiotic therapy, while the American Association of Thoracic Surgery suggests at least two weeks following source control. However, these recommendations are based largely on expert opinion rather than high-quality evidence. Our clinical experience suggests that infectious disease consultation often leads to prolonged antibiotic durations, especially in MDR and tubercular empyema cases. While this approach may reduce recurrence rates, it also carries the risks of adverse drug reactions, increased costs, and the further promotion of antimicrobial resistance. This is particularly concerning in resource-limited settings like Pakistan, where resistance is already a major public health challenge.

The changing microbiological profile of empyema further complicates management. Historically dominated by Gram-positive organisms, the introduction of antibiotics has shifted the burden toward Gram-negative pathogens, many of which exhibit drug resistance. In tubercular empyema, the emergence of MDR-TB presents additional hurdles in both diagnosis and treatment. These microbiological trends highlight the importance of tailored antibiotic and antitubercular regimens informed by culture and sensitivity data. Furthermore, the role of intrapleural fibrinolytics and other adjunctive therapies warrants exploration in our setting, particularly for non-surgical cases.

This study aims to assess the prevalence of multidrug-resistant (MDR) bacterial pathogens and tuberculosis (TB) in patients with empyema requiring surgical intervention. In addition, it seeks to investigate the effectiveness of both thoracoscopic and open decortication techniques in the management of complicated and refractory empyema. By evaluating the microbiological profile and comparing surgical outcomes, the study aims to guide optimal treatment strategies for this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pleural empyema based on clinical, radiological, and microbiological confirmation.
* Patients who underwent surgical decortication for complicated or refractory empyema.

Exclusion Criteria:

* Patients with non-infectious pleural effusions (e.g., malignant pleural effusion, hemothorax, or chylothorax).
* Empyema cases resolved with medical management alone (antibiotics and/or chest tube drainage) without requiring surgical intervention.
* Patients with severe systemic conditions (e.g., end-stage organ failure, terminal malignancy) where empyema management was not the primary therapeutic focus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pleural empyema (MDR bacterial and tuberculous) who underwent surgical decortication (VATS or open thoracotomy) and admitted in thoracic surgery unit of Services hospital Lahore.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
expansion of lung | post-operative day 03 and day 30.
  After decortication, complete re-expansion is defined as ≥90% of the ipsilateral hemithorax occupied by aerated lung on standardized postero-anterior chest radiograph, assessed at full inspiration. Results will be reported as the proportion of participants meeting the ≥90% threshold and units of measurement is percent of hemithorax.

SECONDARY OUTCOMES:
Post-operative pain | post-operative day 01, day 3, day 07 and day 30
  Pain will be assessed using a Visual Analogue Scale (VAS, 0-10 cm), where 0 = no pain and 10 = worst imaginable pain. Assessments will be performed at rest and during deep inspiration/cough. Scores will be collected by trained nursing staff once daily. The primary analysis will report mean VAS score at each time point (with SD).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, Professor of Thoracic Surgery, Principal Investigator — Services Hospital, Lahore
Locations (1):
- Services Institute of Medical Sciences (SIMS), Services Hospital, Lahore, Lahore, Punjab Province, Pakistan